CLINICAL TRIAL: NCT01440231
Title: A Phase II, Multi-Center, Randomized, Double-Blind, Placebo-Controlled, Multidose, 24-Week Dose-Response Study to Evaluate the Efficacy and Safety of Atacicept in Subjects With Systemic Lupus Erythematosus (SLE)
Brief Title: Atacicept Demonstrating Dose RESponSe
Acronym: ADDRESS
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Sponsor: EMD Serono (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EMR 700461-018; BB-IND 11,584 (Other: CDER)
Record Dates: First submitted 2011-09-22; First posted 2011-09-26 (Estimated); Last update posted 2013-08-21 (Estimated); Status verified 2013-08

CONDITIONS: Systemic Lupus Erythematosus
Keywords: Rheumatology; Double-Blind; Placebo-Controlled; Multidose; Dose-Response; Phase II; Systemic Lupus Erythematosus; SLE; Atacicept
MeSH Terms: conditions — Lupus Erythematosus, Systemic | interventions — TACI receptor-IgG Fc fragment fusion protein

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- Arm 1 (Placebo Comparator)
  Interventions: Drug: Placebo
- Arm 2 (Experimental)
  Interventions: Drug: Atacicept
- Arm 3 (Experimental)
  Interventions: Drug: Atacicept
- Arm 4 (Experimental)
  Interventions: Drug: Atacicept
- Arm 5 (Experimental)
  Interventions: Drug: Atacicept

INTERVENTIONS:
Drug: Placebo — Matching placebo administered by subcutaneous injection, once weekly
  Arms: Arm 1
Drug: Atacicept — Atacicept 5 mg administered by subcutaneous injection, once weekly
  Arms: Arm 2
Drug: Atacicept — Atacicept 25 mg administered by subcutaneous injection, once weekly
  Arms: Arm 3
Drug: Atacicept — Atacicept 75 mg administered by subcutaneous injection, once weekly
  Arms: Arm 4
Drug: Atacicept — Atacicept 115 mg administered by subcutaneous injection, once weekly
  Arms: Arm 5

SUMMARY:
Systemic lupus erythematosis (SLE) is an autoimmune disease, meaning that the body's immune system attacks its own organs and tissues. Within the immune system, B-cells and plasma cells make proteins called antibodies, which in autoimmune disease can bind to one's own tissues and are thus referred to as autoantibodies. Atacicept blocks 2 factors in the body, called BLyS and APRIL, which are important for the maintenance of B-cells and plasma cells, and thus the production of antibodies. This study will assess whether treatment with atacicept can reduce SLE disease activity. Atacicept is still an experimental drug, meaning that it is not available outside of a clinical trial, and that its potential benefits and risks have not been fully determined.

A total of 175 subjects are planned to be randomized (35 subjects per treatment arm) in a 1:1:1:1:1 ratio to receive either atacicept 5 mg, atacicept 25 mg, atacicept 75 mg, atacicept 115 mg or matching placebo, given subcutaneously once weekly for 24 weeks.

The primary objective of the trial is to evaluate the efficacy of atacicept compared to placebo in reducing SLE disease activity in subjects treated with standard of care (SoC) therapy and to investigate the dose-response relationship.

The secondary objectives of the trial are:

* To evaluate the effect of atacicept in reducing corticosteroid usage
* To evaluate the safety and tolerability profile of atacicept in subjects with SLE
* To confirm the PK and PD profiles of atacicept in SLE subjects
* To evaluate the changes in the Medical Outcomes Study Short Form General Health Survey [SF-36].

ELIGIBILITY:
Inclusion Criteria:

* Male or female of ≥18 years of age
* Written informed consent
* Diagnosis of SLE satisfying at least 4 out of the 11 ACR criteria during the course of their illness
* Disease duration of at least 6 months
* SLEDAI-2K score ≥ 6 at screening
* Positive test results for antinuclear antibody (ANA) (HEp-2 ANA ≥1:80) and/or anti-double-stranded deoxyribonucleic acid (dsDNA) (≥30 IU/mL) at screening
* Negative serum pregnancy test and highly effective method of contraception for woman of childbearing potential.

Exclusion Criteria:

* Increase in dosing of corticosteroids within 2 weeks prior to screening
* Introduction of MMF within 3 months prior to TD1 or increase in dosing within 1 month before screening
* Change in dosing of immunosuppressants or corticosteroids during the screening period
* Serum IgG < 6g/L
* Estimated Glomerular Filtration Rate (GFR) <50 mL/min/1.73m²
* Urinary protein:creatinine ratio >2 mg/mg
* History of demyelinating disease
* Breastfeeding or pregnancy
* Legal or limited legal capacity

Additional exclusion criteria also apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2012-02; Primary Completion 2013-08 (Estimated); Study Completion 2014-02 (Estimated)

PRIMARY OUTCOMES:
Change from baseline (trial day 1) in SLEDAI-2K Responder Index-50 (SRI-50) at week 24 of therapy | 24 weeks
  The SRI-50 is a modification of the SLEDAI-2K, and allows detection of partial improvements (at least 50%) in SLE signs and symptoms assessed by SLEDAI-2K (Systemic Lupus Erythamtosus Disease Activity Index- 2000).

SECONDARY OUTCOMES:
Change from baseline to Week 24 in corticosteroid dose | 24 weeks
Change from baseline in serum Complement C3 levels at week 24 in subjects with low C3 at baseline | 24 weeks
Change from baseline in serum Complement C4 levels at week 24 in subjects with low C4 at baseline | 24 weeks
Change from baseline in anti-dsDNA antibodies (in subjects with anti dsDNA ≥30 IU/mL at baseline) and in ANA levels (in subjects with HEp-2 ANA ≥1:80 at baseline) at week 24 | 24 weeks
Change from baseline in levels of total Ig and Ig classes (IgG, IgA, and IgM) at week 24 | 24 weekls
The nature (preferred terms) and incidence of AEs | 24 weeks
  Frequency tables summarizing the observed number of AEs by System Organ Class (SOC) and preferred term will be presented per regimen

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Wax, MD, PhD, Study Director — EMD Serono, Senior Medical Director, Rheumatology